CLINICAL TRIAL: NCT04525079
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Parallel Group, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of CT-P59 in Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability and Pharmacokinetics of CT-P59 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Screening
Other Study IDs: CT-P59 1.1; 2020-003065-19 (EudraCT Number)
Record Dates: First submitted 2020-07-30; First posted 2020-08-25 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — regdanvimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1 will receive a dose of CT-P59 or matching placebo
  Interventions: Drug: CT-P59; Drug: Placebo
- Cohort 2 (Experimental): Cohort 2 will receive a dose of CT-P59 or matching placebo
  Interventions: Drug: CT-P59; Drug: Placebo
- Cohort 3 (Experimental): Cohort 3 will receive a dose of CT-P59 or matching placebo
  Interventions: Drug: CT-P59; Drug: Placebo
- Cohort 4 (Experimental): Cohort 4 will receive a dose of CT-P59 or matching placebo
  Interventions: Drug: CT-P59; Drug: Placebo

INTERVENTIONS:
Drug: CT-P59 — CT-P59 will be administered
Drug: Placebo — Placebo-matching CT-P59

SUMMARY:
This is a Phase I study that randomized, double-blind, Placebo-controlled, Parallel Group, Single Ascending Dose Study to evaluate Safety, Tolerability and Pharmacokinetics of CT-P59 in Healthy Subjects.

DETAILED DESCRIPTION:
CT-P59 is a monoclonal antibody targeted against SARS-CoV-2 spike RBD as a treatment for SARS CoV 2 infection. CT-P59 is currently being developed by the Sponsor as a potential treatment for SARS-CoV-2 infection. In this study, safety, tolerability, and pharmacokinetics of CT-P59 will be evaluated in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be randomized in this study:

1. Subject is a healthy male or female subject, aged between 19 to 55 years (both inclusive). Health is defined as no clinically relevant abnormalities identified by Investigator's decision based on a detailed medical history, full physical examination, including blood pressure, heart rate, respiratory rate, and body temperature measurements, 12-lead electrocardiogram (ECG) and clinical laboratory tests prior to the study drug administration.
2. Subject is confirmed as negative in SARS-CoV-2 infection test on screening and Day -1 visits.
3. Subject with a body weight of ≥ 50 kg and a body mass index between 18.0 and 29.9 kg/m2 (both inclusive).
4. Subject is able to understand and to comply with protocol requirements, instructions, and restrictions.
5. Subject voluntarily agrees to participate in this study and has given a written informed consent prior to undergoing any of the screening procedures.

Exclusion Criteria:

Subject meeting any of the following criteria will be excluded from the study:

1. Subject has a medical history or current presence of disease including one or more of the following(s):

   1. History of or current allergic reaction such as asthma, urticaria, angioedema, and eczematous dermatitis considered as clinically significant in the Investigator's opinion or hypersensitivity including known or suspected clinically relevant drug hypersensitivity to any monoclonal antibody or any component of study drug
   2. History of or current medical condition including gastrointestinal, renal, endocrine, neurologic, autoimmune, hepatic, hematological metabolic (including known diabetes mellitus), cardiovascular, or psychiatric condition classed as clinically significant by the Investigator
   3. History of or any concomitant active malignancy
   4. History of or current infection with human immunodeficiency, syphilis, hepatitis B or hepatitis C
   5. History of or current infection requiring a course of systemic anti-infective that was completed within 28 days prior to the study drug administration or a serious infection (associated with hospitalization or which required IV antibiotics) within 6 months before the study drug administration
   6. History of an illness within 28 days prior to the study drug administration that is identified as clinically significant by the Investigator or requires hospitalization
   7. History of surgical intervention or an operation within 28 days prior to the study drug administration or plans to have a surgical procedure during the study period
2. Subject had a history of or concurrent use of medications including any prior therapy of following(s):

   1. Prescription medication (excluding hormonal birth control), over-the-counter drug, dietary supplements or herbal remedies within 7 days or 5 half-lives (whichever is longer) prior to the study drug administration
   2. Any vaccination within 4 weeks prior to the study drug administration
   3. Treatment with any monoclonal antibody, fusion protein, or blood transfusion within 6 months or 5 half lives (which is longer) prior to the study drug administration or current use of biologics
   4. Treatment with any other investigational drug within 6 months or 5 half lives (which is longer) prior to the study drug administration

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-18 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

REFERENCES:
- [Derived] Kim JY, Jang YR, Hong JH, Jung JG, Park JH, Streinu-Cercel A, Streinu-Cercel A, Sandulescu O, Lee SJ, Kim SH, Jung NH, Lee SG, Park JE, Kim MK, Jeon DB, Lee YJ, Kim BS, Lee YM, Kim YS. Safety, Virologic Efficacy, and Pharmacokinetics of CT-P59, a Neutralizing Monoclonal Antibody Against SARS-CoV-2 Spike Receptor-Binding Protein: Two Randomized, Placebo-Controlled, Phase I Studies in Healthy Individuals and Patients With Mild SARS-CoV-2 Infection. Clin Ther. 2021 Oct;43(10):1706-1727. doi: 10.1016/j.clinthera.2021.08.009. Epub 2021 Aug 23. PMID 34551869
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P59 10 mg/kg: Healthy volunteers were administered CT-P59 (10 mg/kg) by intravenously on Day 1. Single-dose was administered to the subjects and monitor up to Day 90.
- CT-P59 20 mg/kg: Healthy volunteers were administered CT-P59 (20 mg/kg) by intravenously on Day 1. Single-dose was administered to the subjects and monitor up to Day 90.
- CT-P59 40 mg/kg: Healthy volunteers were administered CT-P59 (40 mg/kg) by intravenously on Day 1. Single-dose was administered to the subjects and monitor up to Day 90.
- CT-P59 80 mg/kg: Healthy volunteers were administered CT-P59 (80 mg/kg) by intravenously on Day 1. Single-dose was administered to the subjects and monitor up to Day 90.
- Placebo: Healthy volunteers were administered Placebo by intravenously on Day 1. Single-dose was administered to the subjects and monitor up to Day 90.
Period: Overall Study
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 33.5 [21 to 43] | 23.5 [22 to 38] | 28.5 [20 to 34] | 21.5 [19 to 28] | 25 [19 to 43] | 24 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 8 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 8 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 6 | 6 | 6 | 6 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Preliminary Safety and Tolerability of CT-P59
Description: A TEAE includes any untoward medical occurrence in a subject after administration of a study drug, which does not necessarily have to have a causal relationship with this the study drug.
Time Frame: Up to Day 14 after the subject administered with the study drug (Day 1)
Population: Safety set: All subjects who receive a full or partial dose of the study drugs
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | 0 | 2 | 1 | 0 | 1
  Number of Participants with Treatment-Emergent Serious Adverse Events (TESAEs) | 0 | 0 | 0 | 0 | 0
  Number of Participants with Treatment-Emergent Adverse Events of Special Interest (TEAESI) | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Additional Safety of CT-P59 Including Immunogenicity
Description: as for outcome 1
Time Frame: Up to 90 Days
Population: Safety set: All subjects who receive a full or partial dose of the study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | 0 | 4 | 3 | 0 | 1
  Number of Participants with Treatment-Emergent Serious Adverse Events (TESAEs) | 0 | 1 | 0 | 0 | 0
  Number of Participants with Treatment-Emergent Adverse Events of Special Interest (TEAESI) | 0 | 0 | 0 | 0 | 1
  Number of Participants with Anti-Drug Antibody (ADA) positive to CT-P59 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic (PK) Parameters: AUC0-inf and AUC0-last
Description: Data contain Area under the serum concentration-time curve (AUC) from time zero to infinity (AUC0-inf) and Area under the serum concentration-time curve from time zero to the last quantifiable concentration (AUC0-last) of CT-P59.
Time Frame: Up to 90 Days
Population: Pharmacokinetic (PK) set: All subjects who receive a full dose of CT-P59 and have at least 1 evaluable post-treatment PK concentration result
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hr*ng/mL
  Area under the concentration-time curve from time zero to infinity (AUC0-inf) of CT-P59 | 52469185.0 (20377788.54) | 88353384.1 (17775504.91) | 167086786.9 (21899708.77) | 335692549.3 (58444099.42)
  Area under the concentration-time curve from time 0 to the last measured concentration (AUC0-last) | 49593090.2 (15304853.54) | 86246911.1 (15738302.53) | 164581603.9 (21359705.90) | 321167775.4 (47167390.53)

4. Secondary Outcome: Pharmacokinetic (PK) Parameters: AUC0-inf/Dose and AUC0-last/Dose
Description: Data contain Dose normalized AUC0-inf (AUC0-inf/Dose) and Dose normalized AUC0-last (AUC0-last/Dose)
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL/mg
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hr*ng/mL/mg
  Dose normalized AUC0-inf (AUC0-inf/Dose) of CT-P59 (normalized to total body dose) | 68774.1 (22010.25) | 70620.6 (20122.52) | 54763.5 (6031.16) | 58981.8 (7971.33)
  Dose normalized AUC0-last (AUC0-last/Dose) of CT-P59 (normalized to total body dose) | 65200.8 (15941.77) | 68847.6 (18138.86) | 53932.1 (5721.21) | 56474.7 (6274.98)

5. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax
Description: Data contains Maximum observed serum concentration(Cmax) of CT-P59
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 233166.7 (37796.38) | 406333.3 (43647.07) | 1020000.0 (240084.15) | 1941666.7 (267538.16)

6. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax/Dose
Description: Data contains Dose normalized Cmax(normalized to total body dose)(Cmax/Dose) of CT-P59
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL/mg | 307.1 (27.11) | 321.5 (45.42) | 337.0 (91.60) | 342.0 (44.74)

7. Secondary Outcome: Pharmacokinetic (PK) Parameter: Tmax
Description: Data indicates Time to Cmax(Tmax) of CT-P59
Time Frame: Up to 90 Days
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hr | 2.080 [1.57 to 2.6] | 1.575 [1.48 to 5.48] | 2.070 [1.5 to 2.67] | 2.430 [1.53 to 13.63]

8. Secondary Outcome: Pharmacokinetic (PK) Parameter: t1/2
Description: Data contains Terminal half-life (t1/2) of CT-P59
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hr | 473.3 (181.26) | 426.4 (84.52) | 398.6 (36.30) | 526.8 (106.62)

9. Secondary Outcome: Pharmacokinetic (PK) Parameter: %AUCext
Description: Data contains Percentage of AUC0-inf obtained by extrapolation (%AUCext) of CT-P59
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of AUC0-inf
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of AUC0-inf | 3.834 (5.2035) | 2.120 (1.6724) | 1.478 (0.59770) | 4.005 (2.3526)

10. Secondary Outcome: Pharmacokinetic (PK) Parameter: λz
Description: Data contains Terminal elimination rate constant (λz) of CT-P59
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
1/hr | 0.001586 (0.00038316) | 0.001673 (0.00028913) | 0.001751 (0.00016119) | 0.001356 (0.00024242)

11. Secondary Outcome: Pharmacokinetic (PK) Parameter: CL
Description: Data contains Total body clearance (CL) of CT-P59
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL/hr | 15.46 (3.5045) | 14.98 (3.6165) | 18.46 (2.1285) | 17.20 (2.2033)

12. Secondary Outcome: Pharmacokinetic (PK) Parameter: Vz
Description: Data contains Volume of distribution during the elimination phase (Vz) of CT-P59
Time Frame: Up to Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL | 9848.9 (950.01) | 8880.3 (907.10) | 10532.2 (580.96) | 12805.5 (937.08)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the patient signed the ICF until end of study visit (up to Day 90).
Description: From ICF signed date to end of study visit
Arm/Group | CT-P59 10 mg/kg | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 4/6 | 3/6 | 0/6 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P59 10 mg/kg (N=6) | CT-P59 20 mg/kg (N=6) | CT-P59 40 mg/kg (N=6) | CT-P59 80 mg/kg (N=6) | Placebo (N=8)
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P59 10 mg/kg (N=6) | CT-P59 20 mg/kg (N=6) | CT-P59 40 mg/kg (N=6) | CT-P59 80 mg/kg (N=6) | Placebo (N=8)
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04525079/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT04525079/SAP_001.pdf